CLINICAL TRIAL: NCT06614075
Title: The Relationship Between Sociodemographic Characteristics, Lifestyle, and Diet Quality With Diabetes Risk in Overweight and Obese Adults
Brief Title: Diet Quality and Diabetes Risk in Overweight and Obese Adults
Status: Completed | Type: Observational
Sponsor: Ankara Yildirim Beyazıt University (Other)
Responsible Party: Principal Investigator, Rahime Evra KARAKAYA, Principal Investigator, Ankara Yildirim Beyazıt University
Other Study IDs: AnkaraYBU-KARAKAYA002
Record Dates: First submitted 2024-09-20; First posted 2024-09-26 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-09

CONDITIONS: Overweight; Obesity
Keywords: diabetes mellitus; obesity; diet
MeSH Terms: conditions — Overweight; Obesity; Diabetes Mellitus | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adults: Overweight and obese adults
  Interventions: Behavioral: Questionnaire and anthropometric measurement

INTERVENTIONS:
Behavioral: Questionnaire and anthropometric measurement — Questionnaire including sociodemographic characteristics, lifestyle habits, body weight, height, dietary assessment and diabetes risk; Anthropometric measurement including waist circumference

SUMMARY:
The goal of this observational study is to learn about the relationship between diabetes risk with sociodemographic characteristics, lifestyle and diet quality in overweight and obese individuals. The main question it aims to answer is:

Is there a relationship between diabetes risk and diet quality in overweight and obese individuals?

Participants who are overweight and obese will answer survey questions about sociodemographic characteristics and lifestyle behaviors. 24 hour dietary recalls will be taken to evaluate diet quality. FINDRISC questionnaire will be applied to assess diabetes risk.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) ≥25 kg/m²

Exclusion Criteria:

* Diabetes mellitus
* Psychiatric disorders
* Pregnant and lactating

Ages: 19 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Community sample in Ankara, Turkey
Sampling Method: Non-Probability Sample
Enrollment: 1840 (Actual)
Dates: Start 2024-01-15 (Actual); Primary Completion 2024-06-15 (Actual); Study Completion 2024-06-15 (Actual)

PRIMARY OUTCOMES:
Finnish Diabetes Risk Score (FINDRISC) | Baseline
  Scores can range from a minimum of 0 to a maximum of 26 points. According to the FINDRISC scoring system, scores are classified as follows: a score of less than 7 indicates low risk, 7-11 indicates mild risk, 12-14 indicates moderate risk, 15-20 indicates high risk, and a score of less than 20 indicates very high risk.
Healthy eating index-2015 (HEI-2015) | Baseline
  A 24 hour dietary recall was used to assess dietary intake. Nutrient intake obtained from dietary recalls were evaluated using Ebispro for Windows, Stuttgart, Germany; Turkish Version (BeBiS 9). The HEI- 2015 and its sub-scores are calculated based on the quantity of food and nutrient intake per 1,000 kilocalories consumed by individuals. HEI-2015 scores range from a minimum of 0 to a maximum of 100. Based on the calculated scores, a score greater than 80 indicates good diet quality, a score between 51 and 80 is categorized as moderate diet quality, and a score of 50 or less is defined as poor diet quality.

SECONDARY OUTCOMES:
Sociodemographic characteristics | Baseline
  number and percentage
Lifestyle habits | Baseline
  number and percentage
Body weight | Baseline
  Body weight in kg
Height | Baseline
  Height in cm
Waist circumference | Baseline
  waist circumference in cm

CONTACTS AND LOCATIONS:
Overall Officials: Rahime E Karakaya, PhD, Principal Investigator — Ankara Yildirim Beyazıt University
Locations (1):
- Ankara Yıldırım Beyazıt University, Ankara, Çubuk, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Karakaya RE, Elibol E. The relationship between sociodemographic characteristics, lifestyle, and diet quality with diabetes risk in overweight and obese Turkish adults. BMC Public Health. 2025 Jan 2;25(1):5. doi: 10.1186/s12889-024-21248-4. PMID 39748361